CLINICAL TRIAL: NCT03958435
Title: Real-world Retrospective Data Analysis of Adjuvant Therapy for Patients With Stage II-III Colon Cancer After Radical Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: REDUCE201809
Record Dates: First submitted 2018-12-25; First posted 2019-05-22 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-05

CONDITIONS: Stage II Colon Cancer; Stage III Colon Cancer; Adjuvant Therapy
Keywords: Current status; Chemotherapy regimen; Chemotherapy time; Efficacy; Safety; Adjuvant therapy; Stage II-III colon cancer; RWS(Real World Study)
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background:

1. . The incidence and mortality of colon cancer are high in China and in the world.
2. . The treatment of many patients in the real world is not standardized, and there are problems such as over-treatment or under-treatment. To explore the adjuvant treatment of colon cancer in the Chinese population, this study will retrospectively analyze real-world data on adjuvant therapy for colon cancer in Chinese patients after radical surgery.

The purpose of research:

1. . Current status of adjuvant therapy for stage II-III colon cancer in the real world: chemotherapy regimen, chemotherapy time, efficacy, safety, etc.
2. . Comparison of efficacy and safety of different adjuvant chemotherapy time (<3 months vs. >=3 months) in high-risk stage II and III colon cancer patients in the real world
3. . Comparison of efficacy and safety of different adjuvant chemotherapy regimens (XELOX vs. FOLFOX) in high-risk stage II and III colon cancer patients in the real world

ELIGIBILITY:
Inclusion Criteria:

* Patients who are sick after January 2010
* Age is older than 18
* Surgical pathology confirmed TNM stage II-III (AJCC 7th edition) colon cancer

Exclusion Criteria:

* Combine other tumors
* Pathological information is not clear
* Researchers believe that other reasons are not suitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20000 patients diagnosed with stage II-III colon cancer and undergo radical surgery since January 2010.
  The demographic analysis of this study will include but limited in：
  * Demographic characteristics (age, gender, height, weight),
  * Clinical information (Site, TNM(Tumor, regional lymph Node, Metastasis) staging, CEA(Carcinoembryonic Antigen), imaging findings, patient ECOG(Eastern Cooperative Oncology Group)score, PS(Performance Status) score),
  * Pathology information (MMR(Mismatch Repair) status, RAS status, BRAF status, HER2 status, Lymph node, Number of detections, Nerve infiltration, Vascular invasion, Histological type, etc.)
Sampling Method: Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with chemotherapy regimen for adjuvant therapy after stage II and stage III colon cancer | From patients after stage II and stage III colon cancer radical resection to until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months.
  Percentage of patients with chemotherapy regimen for adjuvant therapy after stage II and stage III colon cancer
Percentage of patients with different chemotherapy time for adjuvant therapy for stage II and stage III colon cancer | From patients after stage II and stage III colon cancer radical resection to until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months.
  Percentage of patients with different chemotherapy time for adjuvant therapy for stage II and stage III colon cancer
Percentage of Participants with treatment-related Adverse Events as Assessed by CTCAE v4.0 for adjuvant therapy for stage II and stage III colon cancer | From patients after stage II and stage III colon cancer radical resection to until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months.
  Percentage of Participants with treatment-related Adverse Events as Assessed by CTCAE v4.0 for adjuvant therapy for stage II and stage III colon cancer

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Jiangsu Province People Hospital, Nanjing, Jiangsu
  - Changhai Hospital of Shanghai, Shanghai, Shanghai Municipality
  - SAHZU, Hangzhou, Zhejinag

IPD SHARING:
Plan to Share IPD: Yes